CLINICAL TRIAL: NCT07363174
Title: The Clinical Role of Anogenital Distance in Predicting Pelvic Floor Training Outcomes for Stress Urinary Incontinence
Brief Title: The Clinical Role of Anogenital Distance
Acronym: AGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cigdem Cinar (Other)
Responsible Party: Sponsor-Investigator, Cigdem Cinar, Associate professor doctor, Biruni University
Organization: Biruni University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-KAEK-80-23-51
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Floor Muscle Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelvic Floor Training Outcomes for Stress Urinary Incontinence (Other): All participants will be given pelvic floor muscle strengthening exercises. After 3 months, they will be divided into two groups: those who benefited from the exercises and those who did not.
  Interventions: Other: Anogenital Distance Measurements; Other: pelvic floor muscle strengthening exercises

INTERVENTIONS:
Other: Anogenital Distance Measurements — All anogenital distance (AGD) parameters were measured with participants in the lithotomy position, with the legs positioned at approximately 45°, during the Valsalva maneuver. Measurements were conducted in accordance with standardized protocols to ensure accuracy and reproducibility (6). A stainless-steel digital caliper (VWR® International, LLC, West Chester, PA, USA) was used for all assessments. After each use, the caliper was cleaned with soapy water and disinfected with a 2% alcohol-based chlorhexidine solution.
  Two AGD parameters were recorded: the distance from the anus to the clitoris (AGDAC) and the distance from the anus to the posterior fourchette (AGDAF). In addition, the genital hiatus (GH) was measured from the center of the urethral meatus to the posterior hymenal rim or the perineal midline. To minimize measurement error, all evaluations were performed by the same experienced gynecologist on three separate occasions, and the mean value was used as the final estimate.
Other: pelvic floor muscle strengthening exercises — Following AGD assessment, all patients underwent a standardized pelvic floor muscle training program. Kegel exercises were instructed and supervised by physiatrists with more than ten years of clinical experience in pelvic rehabilitation.
  Before initiating the exercise program, it was essential to confirm that patients could correctly identify and contract their pelvic floor muscles. To achieve this, patients were instructed in Kegel exercises over five consecutive days, performing three sets per day, each set consisting of 8-12 contractions with each contraction lasting 8-10 seconds. Following this initial training, patients were advised to perform the exercises three times daily for a period of three months.
  During monthly outpatient follow-up visits, adherence to the exercise regimen was assessed, and the correctness of the performed exercises was verified. Patients who were unable to perform the exercises correctly received additional instruction.
  Pelvic floor strengthening exercis

SUMMARY:
Aims:

To evaluate the predictive value of anogenital distance (AGD) measurements, including the anus-to-clitoris distance (AGDAC) and genital hiatus (GH), on the success of pelvic floor muscle training (PFMT) in women with stress urinary incontinence (SUI).

Methods:

This cross-sectional, case-control study included 150 adult women with clinically confirmed stress urinary incontinence who completed a three-month PFMT program. All patients' demographic data were recorded, and the anogenital distance (AGDAC, AGDAF) and genital hiatus (GH) were measured using a digital caliper in the lithotomy position. All participants performed supervised Kegel exercises three times daily with monthly follow-up to ensure proper technique and compliance. Patients were then classified as responders or non-responders based on clinical improvement. Associations between PFMT outcomes and AGD parameters, BMI, parity, and other demographic factors were analyzed. All patients will be assessed using the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) before and after treatment.

DETAILED DESCRIPTION:
Clinical and demographic data, including age, weight, height, body mass index (BMI), and number of births, were recorded for all patients at baseline.

All anogenital distance (AGD) parameters were measured with participants in the lithotomy position, with the legs positioned at approximately 45°, during the Valsalva maneuver. Measurements were conducted in accordance with standardized protocols to ensure accuracy and reproducibility (6). A stainless-steel digital caliper (VWR® International, LLC, West Chester, PA, USA) was used for all assessments. After each use, the caliper was cleaned with soapy water and disinfected with a 2% alcohol-based chlorhexidine solution.

Two AGD parameters were recorded: the distance from the anus to the clitoris (AGDAC) and the distance from the anus to the posterior fourchette (AGDAF). In addition, the genital hiatus (GH) was measured from the center of the urethral meatus to the posterior hymenal rim or the perineal midline. To minimize measurement error, all evaluations were performed by the same experienced gynecologist on three separate occasions, and the mean value was used as the final estimate. All patients will be assessed using the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older with confirmed SUI diagnosis who agreed to participate in a 12 weeks pelvic floor rehabilitation program were included in the study

Exclusion Criteria:

* (1) Current pregnancy, (2) history of urinary tract or kidney infection within the last four weeks, (3) diagnosis of diabetes mellitus, (4) previous surgical intervention due to urinary incontinence, (5) known psychiatric disorders, (6) neuromuscular disease, (7) presence of genitourinary fistula, (8) active urogenital malignancy, (9) permanent urinary catheter use, (10) failure to comply with the prescribed exercise program or (11) Pelvic Organ Prolapse Quantification System (POP-Q) Stage 2 (including asymptomatic cases) and above.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
anogenital distance (AGD) parameters | 15 minutes
  Two AGD parameters were recorded: the distance from the anus to the clitoris (AGDAC) and the distance from the anus to the posterior fourchette (AGDAF). In addition, the genital hiatus (GH) was measured from the center of the urethral meatus to the posterior hymenal rim or the perineal midline. To minimize measurement error, all evaluations were performed by the same experienced gynecologist on three separate occasions, and the mean value was used as the final estimate.
International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF) | 1-2 minutes
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a validated patient-reported outcome measure used to assess the severity and impact of urinary incontinence on quality of life. It consists of four items evaluating the frequency of urinary leakage, the amount of urine lost, and the extent to which incontinence affects daily activities, with total scores ranging from 0 to 21 derived from the first three items, while the fourth item identifies situations in which leakage occurs and aids in incontinence subtype classification but is not included in the total score. Higher scores indicate greater symptom severity, and the questionnaire is sensitive to clinical change, with a reduction of 3-4 points considered clinically meaningful and a score of 0 often defined as complete cure. The ICIQ-UI SF is recommended by the International Continence Society, has been translated and validated in multiple languages including Turkish, and is w

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes